# Study Protocol & Statistical Analysis Plan (SAP)

#### Official Title:

Comparative Assessment of Three-Dimensional Soft and Hard Tissue Changes Following Rapid Maxillary Expansion with Face Mask, Mini Maxillary Protractor, and Modified Splints, Elastics, and Chin Cup Protocols in Patients with Class III Malocclusion: A Prospective Randomized Controlled Clinical Trial

**NCT Number:** 

(To be assigned after registration)

**Document Date:** 

[21.02.2024]

# Funding:

This study was supported by the Scientific Research Projects Coordination of Erciyes University (BAP, project number: ID-TDH 2024-13977)

Principal Investigator:

Assoc. Prof. Dr. Gökhan Çoban Department of Orthodontics, Faculty of Dentistry Erciyes University, Kayseri, Turkey

Sub-Investigator:

Research Assistant Dr. Tuba Ünlü Çiftçi Department of Orthodontics, Faculty of Dentistry Erciyes University, Kayseri, Turkey

# **Study Protocol**

# **Study Type and Design**

Interventional, Randomized Controlled Clinical Trial

Allocation: Randomized

Intervention Model: Parallel Assignment

Masking: None (Open Label)
Primary Purpose: Treatment

# **Study Population**

Growing patients with Class III skeletal malocclusion, aged 9–12 years.

#### Interventions

- 1. Rapid Maxillary Expansion with Face Mask (RME/FM)
- 2. Mini Maxillary Protractor (MMP)
- 3. Modified Splint with Elastics and Chin Cup (Modified SEC III)
- 4. Control Group (archival untreated Class III patients)

### **Primary Outcome Measures**

Change in 3D soft tissue profile (facial convexity, mentolabial angle) from baseline to 9 months. Positional changes of anthropometric soft tissue landmarks.

# **Secondary Outcome Measures**

Change in skeletal parameters (SNA, SNB, ANB, overjet, overbite) from baseline to 9 months. Dentoalveolar changes (incisor inclination, linear distances).

#### **Study Dates**

Start Date: February 21 2024

Primary Completion Date: January 09 2025 Study Completion Date: March 03 2025

#### **Ethics**

Approved by the Clinical Research Ethics Committee of Erciyes University (Approval No: 2024/44, Date: Jan 10, 2024). Approval also obtained from the Turkish Medicines and Medical Devices Agency (E-61749811-000-2961523, No: 2023-213).

# Statistical Analysis Plan (SAP)

#### Official Title:

Comparative Assessment of Three-Dimensional Soft and Hard Tissue Changes Following Rapid Maxillary Expansion with Face Mask, Mini Maxillary Protractor, and Modified Splints, Elastics, and Chin Cup Protocols in Patients with Class III Malocclusion: A Prospective

#### Randomized Controlled Clinical Trial

NCT Number:

(To be assigned after registration)

Document Date: [09.01.2025]

# Funding:

This study was supported by the Scientific Research Projects Coordination of Erciyes University (BAP, project number: ID-TDH 2024-13977)

Principal Investigator: Assoc. Prof. Dr. Gökhan Çoban Department of Orthodontics, Faculty of Dentistry Erciyes University, Kayseri, Turkey

Sub-Investigator:

Research Assistant Dr. Tuba Ünlü Çiftçi Department of Orthodontics, Faculty of Dentistry Erciyes University, Kayseri, Turkey

# Statistical Analysis Plan (SAP)

#### **Software**

SPSS Statistics version 21.0 (IBM Corp., Armonk, NY, USA).

# **Normality Testing**

Shapiro-Wilk test used to evaluate distribution of continuous variables.

# **Between-Group Comparisons**

Parametric variables: One-way ANOVA with post-hoc Tukey's tests.

Non-parametric variables: Kruskal-Wallis test with post-hoc Dunn's or Durbin-Conover tests.

# Within-Group Comparisons (T0 vs T1)

Parametric: Paired samples t-test.

Non-parametric: Wilcoxon signed-rank test.

# **Sex-Based Comparisons**

Independent samples t-test for parametric variables.

Mann–Whitney U test for non-parametric variables.

# **Reliability Testing**

Intra-examiner reproducibility assessed by repeating 10 randomly selected cases at 1-month interval.

Reliability calculated using Intraclass Correlation Coefficient (ICC) and Cronbach's alpha.

# **Level of Significance**

A p-value of <0.05 considered statistically significant.